CLINICAL TRIAL: NCT01623076
Title: Collaboration on Neuroimmunology: Question, Understand, Educate, Restore - The Longitudinal CONQUER Study of Rare Neuroimmunologic Disorders
Brief Title: The Longitudinal CONQUER Study of Rare Neuroimmunologic Disorders
Status: Active, not recruiting | Type: Observational
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Benjamin Greenberg, Director, Neuromyelitis Optica and Transverse Myelitis Program, University of Texas Southwestern Medical Center
Other Study IDs: STU 022012-084
Record Dates: First submitted 2012-06-15; First posted 2012-06-19 (Estimated); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Neuromyelitis Optica; Neuromyelitis Optica Spectrum Disorder; Transverse Myelitis; Optic Neuritis
Keywords: Neuromyelitis Optica; Neuromyelitis Optica Spectrum Disorder; Transverse Myelitis; Optic Neuritis; Biorepository
MeSH Terms: conditions — Neuromyelitis Optica; Myelitis, Transverse; Optic Neuritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Patients will donate serum, plasma, DNA, RNA and white blood cells.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Neuromyelitis Optica Spectrum Disorder: Patients diagnosed with NMOSD based on revised diagnostic criteria. Seronegative, anti-AQP4 seropositive and ant-MOG seropositive patients will be included
- Transverse Myelitis and Optic Neuritis: Patients who have had one demyelinating event, not diagnosed with multiple sclerosis and whom are considered at risk for NMO or NMOSD.
- Healthy Controls: patients without a history of CNS inflammation
- Neuromyelitis Optica: patients diagnosed with NMO

SUMMARY:
This study seeks to determine the biologic causes of inflammation in patients with Transverse Myelitis (TM) Neuromyelitis Optica Spectrum Disorder (NMOSD) and related conditions. While patients will be treated according to decisions with their treating physician, this study will collect data and samples from patients prospectively to gain a better understanding of the disease. We are seeking to understand why some patients respond to medications, while others do not. We also seek to understand what happens biologically, preceding relapses. Gathering these data and samples will allow researchers to identify new ways of diagnosing and treating these diseases. Data and samples will be shared with researchers around the world to support collaborative efforts to treat these conditions.

DETAILED DESCRIPTION:
This study seeks to determine the biologic causes of inflammation in patients with Neuromyelitis Optica (NMO), Transverse Myelitis (TM), optic neuritis (ON), related conditions and healthy controls. While patients will be treated according to decisions with their treating physician, this study will collect data and samples from patients prospectively to gain a better understanding of the disease. We are seeking to understand why some patients respond to medications, while others do not. We also seek to understand what happens biologically, preceding relapses. Gathering these data and samples will allow researchers to identify new ways of diagnosing and treating these diseases. Data and samples will be shared with researchers around the world to support collaborative efforts to treat these conditions.

Patients will agree to share medical records, complete questionnaires and donate samples on a timed basis.

ELIGIBILITY:
Inclusion Criteria:

* Age 6 years or greater
* Male or Female
* Patient or Parent (in the case of a minor) able to give informed consent
* For patients 10 to 17, patient able to assent
* Patient diagnosed with NMO, NMOSD, TM or ON

Exclusion Criteria:

* Unable to maintain scheduled visits
* Patient has known HIV or hepatitis C infection

Min Age: 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients previously diagnosed with Neuromyelitis Optica, Neuromyelitis Optica Spectrum Disorder, Transverse Myelitis and Optic Neuritis will be recruited to take part in a longitudinal study of their disease.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2012-06; Primary Completion 2030-06 (Estimated); Study Completion 2030-06 (Estimated)

PRIMARY OUTCOMES:
Measure change in standard clinical assessments over time | Every study visit
  Standard clinical assessments include: relapse information, level of disability based on EDSS score, high and low contract visual acuity, ambulation index, optical coherence tomography, and MRI, and neurologic/physical exam

SECONDARY OUTCOMES:
Measure change in cognition measures over time | Every study visit
  Cognition measures include the SDMT, JLO, and PASAT
Measure change in self-reported quality of life surveys | Every study visit
  Surveys include MSNQ, MSQOL-54, QIDS, BDI-II, FSS, ESS, MFIS, BPI, and Neuro-QoL
B cell population changes | Up to 5 years
  Measure B cell subtypes and changes over time

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin M Greenberg, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- The University of Texas Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified data can be shared with IRB approved researchers upon request and approval from PI

REFERENCES:
- See also: Transverse Myelitis Association — http://www.myelitis.org/